CLINICAL TRIAL: NCT02395263
Title: Proof Of Concept Study of Yuxintine in the Treatment of Major Depressive Disorder(MDD): a Randomized, Double-Blind, Placebo-Paralleled,Dose-Finding, Multicenter Clinical Trial
Brief Title: Comparison of Yuxintine With Placebo in Treatment of MDD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Innovative Research Center of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Yuxintine Capsule-MDD-Ⅱb; 2012ZX09303-003 (Other Grant/Funding Number: China National Major Project)
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Yuxintine 200mg per day (Experimental): Yuxintine 200mg oral, once a day, 6 weeks
  Interventions: Drug: Yuxintine
- Yuxintine 300mg per day (Experimental): Yuxintine 300mg oral, once a day, 6 weeks
  Interventions: Drug: Yuxintine
- Yuxintine 400mg per day (Experimental): Yuxintine 400mg oral, once a day, 6 weeks
  Interventions: Drug: Yuxintine
- Placebo (Placebo Comparator): Placebo oral, once a day, 6 weeks
  Interventions: Drug: Yuxintine

INTERVENTIONS:
Drug: Yuxintine

SUMMARY:
The purpose of this study is to determine whether Yuxintine Capsule in different doses are effective in the treatment of Depression.

And to explore the preliminary information of safety and efficacy of Yuxintine Capsule in the Chinese Patients with Depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of major depressive disorder(MDD) based on the criteria of DSM-IV-TR, single episode or recurrent episode, not accompanied with psychotic symptoms. Coding of diagnosis included: 296.2 and 296.3.
* The Subject with Heart-Spleen Deficiency based on the CTM.
* The total score of MADRS is ≥22 in both screening visit and baseline visit.
* The total score of HAMD-17 is ≥18 and ≤30, AND item 1 ≥2 in both screening visit and baseline visit.
* The subject understands and consents to takes part in this clinical trials. The subjects should sign informed consent.

Exclusion Criteria:

* The subject made a suicide attempt in recent 6 months or has a score ≥3 on item 3(suicide assessment) of the HAMD.
* The subject has a current DSM-Ⅳ-TR axisⅠpsychiatric diagnosis other than depression.
* When the MADRS score of baseline visit compares with the screening visit, the decreasing rate is ≥25%.
* Any unstable cardiovascular, hepatic, renal, endocrine(thyroid gland dysfunction), blood(e.g. bleeding tendency),or other medical disease.
* Had a history of seizure disorder,except infantile febrile convulsion.
* The subject has accepted psychosurgery or electroconvulsive therapy within 3 months.
* With psychotic symptoms.
* The subject has a history of mania episode, including manic, mixed or rapid cycle attack.
* The subject has a current diagnosis or history of depression due to any other psychotic disorder or a general medical condition.
* The subject with refractory depressive disorder,i.e.the patients who used at least two different mechanisms antidepressants with adequate dosage and duration treatment still had no respond.
* Clinically significant electrocardiographic(ECG) abnormalities or abnormal laboratory values(eg. Hepatic function above 1.5 times of clinical toplimit, renal function index above toplimit, abnormal coagulation function and clinical significance of abnormality, i.e. Prothrombin time shorten or extend more than 3 seconds or a dynamic variation or APTT prolonged more than 10 seconds,AND fibrinogen L or been progressive decline, or > 4.0 g/L).
* The subject has a diagnosis of alcohol or other substance abuse or dependence at least 1 years prior to the baseline visit.
* Known hypersensitivity to Ginseng, or at least to two kinds of drugs, or serious allergic physique.
* Women who were pregnant, breast-feeding, or planning to become pregnant during study. Men who have request to fertility during study period. The subject could not take safe and effective birth control measures.
* The subject could not take medication according to the doctor's advice.
* The subject uses antidepressant drug normally before 2 weeks of screening, and stops using psychotropic drug less than 7 half-life period (monoamine oxidase inhibitor more than 2 weeks).
* The subject has participated in a drug clinical trial within 3 months before screening.
* The investigator think the subject is unsuitable to enrol in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The change of total score from baseline in MADRS scale | 6 weeks

SECONDARY OUTCOMES:
clinical response rate according to MADRS | 6 weeks
clinical remission rate according to MADRS | 6 weeks
CGI(CGI-S,CGI-I) | 6 weeks
The change of total score from baseline in HAMD scale | 6 weeks
decreasing rate from baseline in HAMD scale | 6 weeks
clinical remission rate according to HAMD | 6 weeks
change from baseline in HAMA | 6 weeks
Traditional Chinese Medicine Syndrome Scale | 6 weeks

OTHER OUTCOMES:
vital sign | 6 weeks
  Blood pressure, heart rate, temperature and respiratory rate
The Arizona Sexual Experience Scale (ASEX) | 6 weeks
laboratory examination | 6 weeks
  Blood RT, Urinalysis,Hepatic function,Renal function,FBG,Lipid,Thyroid Function, Blood Coagulation Test and U-HCG
AE(adverse events) | 6 weeks
ECG | 6 weeks
Early Termination | 6 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Shenzhen Mental Health Center, Shenzhen, Guangdong
  - the People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - Hebei Mental Health Center, Shijiazhuang, Hebei
  - Hunan Brain Hospital, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality